CLINICAL TRIAL: NCT00298987
Title: Study of Dasatinib (BMS-354825) in Subjects With Chronic Myelogenous Leukemia With Accelerated or Myeloid or Lymphoid Blast Phase or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Who Are Resistant to or Intolerant of Imatinib Mesylate
Brief Title: A Study of Dasatinib in Patients With Chronic Myelogenous Leukemia Who Are Resistant or Intolerant of Imatinib Mesylate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-033
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2008-06

CONDITIONS: Leukemia, Myeloid, Chronic; Leukemia, Lymphocytic, Acute, L2
Keywords: Chronic Myeloid Leukemia Accelerated and Blast Phase; Leukemia, Acute, Philadelphia-Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Leukemia | interventions — Dasatinib

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 70 mg, Twice daily, 2 months.
  Other Names: Sprycel

SUMMARY:
The purpose of this clinical research study is to provide dasatinib treatment to patients with advanced chronic myelogenous leukemia (CML) or Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL) who no longer can tolerate treatment with imatinib. The safety of the treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of accelerated phase or blast phase CML or Ph+ ALL
* Intolerant or resistant to imatinib mesylate
* 18 years of age or older
* ECOG performance 0-2 (greater than 50% of time out of bed)
* Adequate liver and kidney function

Exclusion Criteria:

* Pregnant or breastfeeding females
* History of significant cardiac disease
* History of significant bleeding disorder (not CML)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Provide therapy to patients for which there is no therapeutic alternative

SECONDARY OUTCOMES:
Safety data collection

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (30):
  - Local Institution, Corona, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Waterford, Connecticut
  - Local Institution, Daytona Beach, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Lawrenceville, Georgia
  - Local Institution, Beach Grove, Indiana
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Iowa City, Iowa
  - Local Institution, Kansas City, Kansas
  - Local Institution, Salina, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Louisville, Kentucky
  - Local Institution, Boston, Massachusetts
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, Detroit, Michigan
  - Local Institution, Santa Fe, New Mexico
  - Local Institution, New York, New York
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Lawton, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Portland, Oregon
  - Local Institution, Providence, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Spokane, Washington
  - Local Institution, Sheboygan, Wisconsin
- Canada (5):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec